CLINICAL TRIAL: NCT05043805
Title: The Study of Risk Factors and Intervention for Children With Chronic Irritability - a Preliminary Approach With Epidemiological, Neuropsychological and Neuroinflammation Studies
Brief Title: Dextromethorphan Added on for Children With Chronic Irritability
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Chin-Bin Yeh, MD, PhD, Principal Investigator, Professor, Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2-108-05-085
Record Dates: First submitted 2021-08-27; First posted 2021-09-14 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Irritable Mood
MeSH Terms: interventions — Dextromethorphan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dextromethorphan (Active Comparator): add on therapy
  Interventions: Drug: Dextromethorphan
- placebo (Placebo Comparator): add on therapy
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Dextromethorphan — add on therapy
  Other Names: regrow
  Arms: Dextromethorphan
Other: placebo — add on therapy
  Arms: placebo

SUMMARY:
Dextromethorphan Added on for Children With Chronic Irritability

DETAILED DESCRIPTION:
Objectives:

It is known that the etiology and mechanism of neuropsychiatric diseases may be related to nerve inflammation. It has been found that dextromethorphan (DM) is an active ingredient in cough-remedies, which can protect neurons in glial cell cultures in the rat brain from inflammatory substances. Although the mechanism of DM is still unknown, it may be related to the regulation of immune dysfunction. Therefore the purpose of this present study was to investigate the adjuvant treatment with DM in the children and adolescents with chronic irritability.

Methods:

This randomized double-blind clinical trial will evaluate 120 outpatients, aged between 7 and 17 years, with chronic irritability. The study subjects will be randomly assigned into one of the two groups: receiving routine medicine plus DM or routine medicine plus placebo for 8 weeks. Assessments comprising the parents' reported Mood Disorder Questionnaire (MDQ), Affective Reactivity Index (ARI), the Chinese version of the Child Behavior Checklist (CBCL-C) scale, the Swanson, Nolan and Pelham Questionnaire (SNAP-IV), the Sleep Disturbance Scale for Children (SDSC), Problematic smartphone use (PSU) and Checklist for Autism Spectrum Disorder-Chinese Version (CASD-C). Comparison will be done between groups at baseline and at 8 weeks before-and-after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 7 to 17 who have irritability symptoms will be recruited. They will be screened for the irritability symptoms with ARI scale.

Exclusion Criteria:

* Patients who are not willing to participate in the study after detailed explanation.
* Patients who could not follow the investigator's instructions.
* Patients who have problems to express questions or emotional problems exactly.
* Patients who have severe neurological or mental illness like epileptic disorder, history of stroke, schizophrenia, bipolar disorder, mental retardation or uncontrolled suicide risk.
* Patients who have severe medical illness or surgical conditions like uncontrolled abnormal thyroid function, history of heart attack, uncontrolled hypertension.
* Patients who are allergic to methylphenidate or dextromethorphan.
* Patients with autoimmune disorders
* Patients with asthma or severe infection disorder currently or in the previous two months to avoid the influence of the level of cytokines.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2021-05-09 (Actual); Primary Completion 2024-04-05 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Irritability severity | 8 weeks
  The investigators will measure if the severity improve after using regrow by the ARI scale.

SECONDARY OUTCOMES:
ADHD severity | 8 weeks
  The investigators will measure if the severity improve after using regrow with regular drug by the SNAP-IV scale.

CONTACTS AND LOCATIONS:
Overall Officials: Chin-Bin Yeh, M.D., Ph.D., Principal Investigator — Tri-Service General Hospital
Locations (1):
- Tri-Service General Hospital, National Defense Medical Center, Taipei, Taiwan